CLINICAL TRIAL: NCT04621890
Title: Behavioral Incentive Meal Dose Engagement in Adolescents With Type 1 Diabetes
Brief Title: HCT Cash-Only INcentive to Promote Mealtime Insulin DOSE Engagement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Sarah Tsai, Pediatric Endocrinologist, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001086
Record Dates: First submitted 2020-10-03; First posted 2020-11-09 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: There will be 3 arms to this study. Two of these will involve behavioral interventions - LOAN2DOSE and COIN2DOSE. The remaining arm will be the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LOAN2DOSE (Experimental): From one-week post-randomization to the 12-week study visit, youth randomized to this treatment arm will receive personalized feedback via monetary deductions from a virtual bank of $210 for missed doses of insulin at mealtimes. According to the methodology for calculating BOLUS(1) breakfast will be 0600-1000, lunch will be 1100-1500, and dinner will be 1600-2000. Thus, we will deduct $0.50 per mealtime with at least one meal-associated (carbohydrate-associated) insulin bolus missed (maximum -$1.50/day). Youth can also lose an additional amount of up to $5.00/week for weeks during which they don't achieve at least 5 days of 3 mealtime insulin boluses. Finally, we will deduct the virtual account up to $2.00 per week for failing to share their insulin use data at least two times per week with the study team during the three-month treatment phase (maximum deduction of $24.00). Maximum total deductions is $210.
  Interventions: Behavioral: LOAN2DOSE and COIN2DOSE
- COIN2DOSE (Experimental): From one-week post-randomization to the 12-week study visit, youth randomized to this treatment arm will receive personalized feedback via monetary incentives for dosing insulin at mealtimes. Mealtimes will be defined based on hour of the day and the presence of a carbohydrate entry associated with the insulin bolus. Breakfast will be 0600-1000, lunch will be 1100-1500, and dinner will be 1600-2000. Thus, we will reimburse youth up to $0.50 per mealtime with at least one meal-associated (carbohydrate-associated) insulin bolus completed (maximum $1.50/day). We will offer the opportunity for youth to earn a bonus reimbursement of up to $5.00/week for weeks during which they achieve at least 5 days of 3 mealtime insulin boluses. Finally, we will pay youth up to $2.00 per week for sharing their insulin use data at least two times per week with the study team during the three-month treatment phase (maximum $24.00). Therefore, maximum total incentive available is $210.
  Interventions: Behavioral: LOAN2DOSE and COIN2DOSE
- Control (No Intervention): This group will engage have usual diabetes care without intervention. They will fill out all questionnaires, attend clinic visits and provide A1C samples at the same times as the participants in the other groups.

INTERVENTIONS:
Behavioral: LOAN2DOSE and COIN2DOSE — This is a behavioral economics intervention designed to help improve meal time bolusing behaviors in youth with type 1 diabetes.
  Arms: COIN2DOSE; LOAN2DOSE

SUMMARY:
Type 1 Diabetes (T1D) is a serious disease that happens because the body cannot control blood glucose (sugar) levels. People with T1D need insulin shots because their body does not make insulin. Insulin lowers blood sugar levels. When blood sugar levels are too high or too low it causes medical problems.

Youth with T1D can really impact their own health if they follow their T1D treatment plan. However, even with the help of doctors, nurses, and family, most adolescents find it hard to follow their diabetes plan close enough to meet their A1C goal. It is very common for adolescents to forget to give an insulin bolus for meals. When insulin doses are missed, there is a greater chance for poor blood sugar control. When adolescents follow their diabetes plan closely, they have better blood sugar control and overall health.

Two behavioral economic interventions will be evaluated. COIN2DOSE (Cash-Only INcentive to promote mealtime insulin DOSE Engagement) and LOAN2DOSE (Behavioral Economic concept that uses an economic loss aversion approach to promote insulin dose engagement in adolescents with Type 1 Diabetes). These programs were designed to improve blood sugar control by decreasing the number of missed mealtime boluses. For COIN2DOSE, we will offer the opportunity for youth to earn a bonus reimbursement during which they achieve at least 5 days of 3 mealtime insulin boluses. Finally, we will pay youth up for sharing their insulin use data at least two times per week with the study team during the three-month treatment phase. For LOAN2DOSE, the participants will start with a monetary "balance" and will keep it if they bolus as instructed - at least 5 days of 3 mealtime insulin boluses. If they do not do this, their balance will decrease throughout the study.

DETAILED DESCRIPTION:
The long-term goal is to develop effective ways to improve glycemic control in youth with T1D. To that end, we propose to specifically evaluate the effectiveness, feasibility, and usability of two new behavioral economic interventions in diabetes care: an automated meal detection and patient engagement device to promote meal-time insulin dosing behavior (AIM2DOSE) and an economic incentive (COIN2DOSE) to promote patient engagement with mealtime insulin dosing behavior. If initially efficacious, our results will serve as the basis for an R01 submission(s) to conduct a fully powered efficacy trial of LOAN2DOSE and COIN2DOSE. This study is significant as omission of mealtime boluses is one of the common reasons for suboptimal diabetes control in youth. This project is highly innovative because it will: 1) target youth who are predicted by artificial intelligence to experience a worsening in glycemic control, 2) use a just-in-time intervention to improve mealtime insulin dosing behavior, and 3) use an economic incentive intervention to improve mealtime insulin dosing behavior.

Study Design The study is an unblinded, 3-arm, randomized, controlled trial. After successful screening and consent, individuals will wear a blinded Dexcom G6 Pro CGM inserted 1 week after consent. . At the baseline visit (visit 1; day 1), participants will be randomized to the LOAN2DOSE, COIN2DOSE, or control treatment arms and will be trained on the procedures appropriate to their treatment arm. Participants will also complete baseline measures by questionnaire. Participants will complete procedures specific to their treatment arm weekly. Visit 2 will occur after 12 weeks (90 days). Participants will stop any treatment interventions after this visit. A1C and questionnaire measures will be completed, and participants will again wear the Dexcom G6 Pro CGM for 10 days (the device will be returned by mail post-visit). Participants will receive no treatment intervention from week 13 to week 24. Participants will return for visit 3 at week 24. Again, A1C and questionnaire measures will be completed and participants will wear the Dexcom G6 Pro CGM for 10 days.

All study participants will also have the option to participate in a focus group discussion (FGD) on general AI ethical issues (control group) or intervention experiences (intervention group).

Parents of children who meet inclusion criteria may also elect to participate in a focus group.

Study Visits Study visits may occur in-person or remotely (i.e., from home). Procedures will be adapted to accommodate both scenarios.

Individuals who have been predicted via an artificial intelligence-intelligence based model to experience a rise in A1C in the near future (90 days) will be approached for recruitment. 36 participants will be recruited from the Children's Mercy Diabetes Center (any clinic or hospital location). Based on preliminary data review of our clinic population, there were at least 81 individuals who met inclusion criteria who were seen in clinic in the month of May 2019 alone. Patients will be randomized to LOAN2DOSE, COIN2DOSE, or control group using a 1:1:1 randomization scheme.

Intervention:

To identify an at-risk population for more intensive intervention opportunities, the Children's Mercy Diabetes Center now routinely uses a validated prediction model based on advanced machine learning (random forest method) and natural language processing to identify individuals who are predicted experience a rise in A1C in the next 90 days. The model analyzes all patients who presented for a diabetes visit in the prior week. To accomplish this task, the complete health record for the CMH Diabetes Center registry is analyzed. We will select patients from this cohort for recruitment into the present study.

COIN2DOSE intervention: From one-week post-randomization to the 12-week study visit, youth randomized to this treatment arm will receive personalized feedback via monetary incentives for dosing insulin at mealtimes. We will define mealtimes based on hour of the day and the presence of a carbohydrate entry associated with the insulin bolus. Breakfast will be 0600-1000, lunch will be 1100-1500, and dinner will be 1600-2000. Thus, we will reimburse youth per mealtime with at least one meal-associated (carbohydrate-associated) insulin bolus completed. We will offer the opportunity for youth to earn a bonus reimbursement for weeks during which they achieve at least 5 days of 3 mealtime insulin boluses. Finally, we will pay youth per week for sharing their insulin use data at least two times per week with the study team during the three-month treatment phase.

LOAN2DOSE intervention: From one-week post-randomization to the 12-week study visit, youth randomized to this treatment arm will receive personalized feedback via monetary deductions from a virtual bank of $210 for missed doses of insulin at mealtimes. We will define mealtimes based on hour of the day and the presence of a carbohydrate entry associated with the insulin bolus. According to the methodology for calculating BOLUS(1) breakfast will be 0600-1000, lunch will be 1100-1500, and dinner will be 1600-2000. Thus, we will deduct $0.50 per mealtime with at least one meal-associated (carbohydrate-associated) insulin bolus missed (maximum -$1.50/day). Youth can also lose an additional amount of up to $5.00/week for weeks during which they don't achieve at least 5 days of 3 mealtime insulin boluses. Finally, we will deduct the virtual account up to $2.00 per week for failing to share their insulin use data at least two times per week with the study team during the three-month treatment phase (maximum deduction of $24.00). Therefore, maximum total deductions is $210.

ELIGIBILITY:
Inclusion Criteria:

* Aged 12-17.99 years
* The youth must have been diagnosed with T1D for at least 6 months
* The youth must have attended at least 2 routine T1D standard of care visits in the past 12 months
* The youth must be using an insulin delivery device capable of recording, storing, and downloading insulin bolus behaviors (insulin pump or smart Bluetooth insulin pen that can be uploaded to standard clinic upload software).
* The youth must have a current A1C >7.2% and/or be predicted to have a rise in A1C in of 0.3% or higher the next 90 days.
* Not pregnant or planning to become pregnant by self-report.

Exclusion Criteria:

* Participants with any type of diabetes mellitus other than T1D
* Participant has any disease causing anemia or affecting red blood cell physiology (which would impact A1C)
* Participant has a physical disability, which in the opinion of the investigator would interfere with individual's ability to feed themselves or use one's hands to facilitate eating
* Participants with no internet access or ability to upload device(s) to data aggregation software that is accessible to study team.

For Focus Groups:

Any parent or legal guardian whose child is eligible for the study is invited to participate in a focus group discussion.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change in A1C (ΔA1C90-day) from baseline visit (visit 1) to 90-day visit (visit 2) | baseline and 90 days
  A1C is a validated indicator of glycemic control.

SECONDARY OUTCOMES:
Change in A1C (ΔA1C180-day) from baseline visit (visit 1) to 180-day visit (visit 3). | baseline and 180 days
  A1C is a validated indicator of glycemic control.
Change in percent time in range 70-180 mg/dL (%TIR70-180) from baseline visit (visit 1) to 90-day visit (visit 2) and to 180-day visit (visit 3). | baseline, 90 and 180 days
  Participants blood sugars will be obtained from Dexcom, insulin pump, glucometer or other device.
Change in percent time hyperglycemic (>180 mg/dL; %Hyper>180) from baseline visit (visit 1) to 90-day visit (visit 2) and to 180-day visit (visit 3). | baseline, 90 and 180 days
  Participants blood sugars will be obtained from Dexcom, insulin pump, glucometer or other device.
Change in percent Time hypoglycemic (<70 mg/dL; %Hypo<70) from baseline visit (visit 1) to 90-day visit (visit 2) and to 180-day visit (visit 3). | baseline, 90 and 180 days
  Participants blood sugars will be obtained from Dexcom, insulin pump, glucometer or other device.
Change in percent Time severely hypoglycemic (<54 mg/dL) (%Hypo<54) from baseline visit (visit 1) to 90-day visit (visit 2) and to 180-day visit (visit 3). | baseline, 90 and 180 days
  Participants blood sugars will be obtained from Dexcom, insulin pump, glucometer or other device.
Change in mealtime insulin BOLUS score (BOLUS) from baseline visit (visit 1) to 90-day visit (visit 2) and to 180-day visit (visit 3). | baseline, 90 and 180 days
  BOLUS (Frequency of mealtime insulin bolusing) score is a validated measure of frequency of meal-time insulin bolusing adherence.
For LOAN2DOSE treatment group, proportion of participants wearing the apple watch throughout the 90-day intervention period >75% of days. | baseline, 90 and 180 days
  For LOAN2DOSE treatment group, proportion of participants wearing the apple watch throughout the 90-day intervention period >75% of days.
For LOAN2DOSE treatment group, proportion of participants who deliver insulin bolus doses within 10 minutes of >75% of mealtime bolus reminders. | baseline, 90 and 180 days
  For LOAN2DOSE treatment group, proportion of participants who deliver insulin bolus doses within 10 minutes of >75% of mealtime bolus reminders.
For LOAN2DOSE treatment group, proportion of participants who complete >90% of study procedures throughout the intervention and post-intervention study procedures. | baseline, 90 and 180 days
  For LOAN2DOSE treatment group, proportion of participants who complete >90% of study procedures throughout the intervention and post-intervention study procedures.
For COIN2DOSE treatment group, proportion of parents who endorse the feasibility of providing an economic incentive equivalent to that used in the intervention. | baseline, 90 and 180 days
  For COIN2DOSE treatment group, proportion of parents who endorse the feasibility of providing an economic incentive equivalent to that used in the intervention.
For COIN2DOSE treatment group, >75% of participants will have a score of at least 14 out of a total possible 18 points on Diabetes Treatment Satisfaction Questionnaire (teen version). | baseline, 90 and 180 days
  Diabetes Treatment Satisfaction Questionnaire (teen version) is a validated measure of satisfaction with personal health care delivery. There are 6 items, with scores ranging from +3 to -3. A higher score indicates greater treatment satisfaction.
Change in trust in provider from baseline visit (visit 1) to 90-day visit (visit 2) and to 180-day visit (visit 3). | baseline, 90 and 180 days
  Trust in provider: Will be measured as a change score (visit 2-visit 1; visit 3-visit 1) with 10-items from the validated Wake Forest Physician Trust Scale. Response categories: Strongly agree, agree, neutral, disagree, and strongly disagree.
Change in perceived involvement in care from baseline visit (visit 1) to 90-day visit (visit 2) and to 180-day visit (visit 3). | baseline, 90 and 180 days
  Will be measured as a change score with 13-items from the Perceived Involvement in Care Scale. Response categories: Strongly agree, somewhat agree, neutral, somewhat disagree, and strongly disagree.
Change in health-related empowerment from baseline visit (visit 1) to 90-day visit (visit 2) and to 180-day visit (visit 3). | baseline, 90 and 180 days
  Will be measured as a change score with 8-items from the Health-related empowerment scale. Response categories: Strongly agree, somewhat agree, neutral, somewhat disagree, and strongly disagree

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Mercy Kansas City, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD at this time.

DOCUMENTS (1):
  • Study Protocol (2023-12-26): https://cdn.clinicaltrials.gov/large-docs/90/NCT04621890/Prot_000.pdf